CLINICAL TRIAL: NCT04096209
Title: The Effect on Dental Implant Stability With and Without Using 1:1 Mixture of Autogenous Bone and Anorganic Bovine Bone Minerals Particulates in Immediate Implant Placement in the Dental Esthetic Zone (A Randomized Clinical Trial)
Brief Title: Immediate Implant Placement in the Esthetic Zone With and Without Using Autogenous Mixed With Xenograft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherine Osama El ebiary, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CairoUimplant 2
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Badly Decayed Teeth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Graft-less and grafting using xenograft and autograft (Experimental): Extraction of badly decayed teeth with immediate implant placement using graft-less and grafting using autogenous bone and xenograft between the implant and labial socket bone
  Interventions: Device: autograft mixed with xenograft bone

INTERVENTIONS:
Device: autograft mixed with xenograft bone — Eligible patients will be randomized in equal proportions between control group (immediate implant placement without bone grafts in the jumping gap) and study group (immediate implant placement with a mixture of Xenograft and autogenous bone placed in the jumping gap).
  All patients will be evaluated by proper history taking and thorough clinical and radio graphical examination and assessed according to the inclusion and exclusion criteria.
  Patients of both groups will be subjected to Cone beam Computed tomography (CBCT).
  Primary impression will be taken, a study model will then be poured and then waxing up will be performed.
  Patients will be instructed to rinse with chlorhexidine 0.1% mouthwash. Articaine 4% (1:100,000) local anesthesia will be given to the patient. Atraumatic extraction of the tooth or remaining root using No. 15c lancet and periotome

SUMMARY:
Xenografts are graft materials derived from the inorganic portion of animal bones; the most common source is bovine the removal of the organic component are processed to remove their antigenicity, while the remaining inorganic components provide a natural matrix as well as an excellent source of calcium. The disadvantage of xenografts is that they are only osteoconductive and the resorption rate of bovine cortical bone is slow.

However leaving the jumping gap empty has been the gold standard for immediate implantation as the formed blood clot will allow bone fill in that area.

DETAILED DESCRIPTION:
Not using a grafting material in the jumping gap was chosen as a comparator as it's the standard procedure usually applied and showed high success rates. This should allow us to assess whether the chosen grafting material would have a positive influence on the study outcomes as compared to it.

Intraoral and extraoral autologous bone grafts could be considered as the "Gold standard" pre-prosthetic dentoalveolar reconstruction of atrophic jaws with cortico-cancellous bone grafts from intraoral and/or extraoral donor sites as a predictable technique for the facilitation of dental rehabilitation of atrophic ridges, associated with high bone survival rate and long term implant success. Autogenous bone corresponds to bone graft obtained from the same individual. It is considered the gold standard for filling of bone defects since it allows (I) osseointegration: direct contact with bone tissue without fibrous tissue ; (II) osteoconduction: support to bone growth (III) osteoinduction: differentiation of mesenchymal cells of surrounding tissue (receptor site) into osteoblastic cells ; and (IV) osteogenesis: bone neoformation by osteoblastic cells present in the graft material. Although few mature osteoblasts survive to grafting, precursor cells are responsible for the osteogenic potential

ELIGIBILITY:
Inclusion Criteria:

* Age from 20-60 years
* Both sexes
* non-restorable maxillary incisors, canine and premolars
* Good oral hygiene
* Adequate bone height apical to the alveolus of the failing tooth

Exclusion Criteria:

* Systematic disease which affect osseointegration (uncontrolled diabetes, cancer, etc...)
* Bad oral hygiene
* Bruxism, clenching, deep bite, edge to edge and abnormal habits
* Non-treated periodontal diseases
* Pregnancy and smokers
* Severe infection
* Absence of labial plate of bone (Fenestration, dehiscence).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 4-6 months
  implant stability will be measured using osstell

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] El Ebiary SO, Atef M, Abdelaziz MS, Khashaba M. Guided immediate implant with and without using a mixture of autogenous and xeno bone grafts in the dental esthetic zone. A randomized clinical trial. BMC Res Notes. 2023 Nov 13;16(1):331. doi: 10.1186/s13104-023-06612-8. PMID 37957760